CLINICAL TRIAL: NCT04243434
Title: An Open-Label, Randomized, Pharmacokinetic Study of vinCRIStine Sulfate LIPOSOME Injection Ready-to-Use (VSLI-RTU) Formulation (1-Vial) and Marqibo® Formulation (3-Vials) in Patients With Hematological Malignancies
Brief Title: PK Study on Ready-to-Use Injection (VSLI-RTU) 1 Vial & 3 Vial Formulation Marqibo® in Hematological Malignant Patients
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Acrotech Biopharma Inc. (Industry)
Collaborators: Axis Clinicals Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SPI-MAR-101
Record Dates: First submitted 2019-10-17; First posted 2020-01-28 (Actual); Last update posted 2020-04-16 (Actual); Status verified 2020-04

CONDITIONS: Hematologic Diseases
Keywords: Hematology; Hematological Malignancy; CHOP; R-CHOP
MeSH Terms: conditions — Hematologic Diseases; Hematologic Neoplasms | interventions — Vincristine; AC protocol; Prednisone; Doxorubicin; R-CHOP protocol; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort A (Experimental): Marqibo formulation given at a dose of 2.25 mg/m2 with no dose cap during Cycle 1, and VSLI-RTU formulation given at 2.25 mg/m2 with no dose cap during Cycle 2.
  Interventions: Drug: Vincristine Sulfate Liposome; Combination Product: CHOP; Combination Product: R-CHOP
- Cohort B (Experimental): VSLI-RTU formulation given at a dose of 2.25 mg/m2 with no dose cap during Cycle 1 and Marqibo formulation given at 2.25 mg/m2 with no dose cap during Cycle 2.
  Interventions: Drug: Vincristine Sulfate Liposome; Combination Product: CHOP; Combination Product: R-CHOP

INTERVENTIONS:
Drug: Vincristine Sulfate Liposome — Eligible patients will be randomized in a 1:1 ratio to one of 2 treatment cohorts (Cohorts A or B) to receive either the first cycle of treatment with the VSLI-RTU formulation or the Marqibo formulation and crossover to the other formulation for the second cycle.
  Other Names: Marqibo
Combination Product: CHOP — CHOP to be administered on Day 1 on Cycle 1 & 2 ( 21-day Cycle) & prednisone administration on Days 2 to 5 on Cycle 1 & 2 ( 21-day Cycle)
  Other Names: cyclophosphamide. doxorubicin, vincristine , and prednisone; Adriamycin, (Oncovin)
Combination Product: R-CHOP — R-CHOP to be administered on Day 1 on Cycle 1 & 2 ( 21-day Cycle) & prednisone administration on Days 2 to 5 on Cycle 1 & 2 ( 21-day Cycle)
  Other Names: cyclophosphamide. doxorubicin, vincristine , prednisone + Rituximab

SUMMARY:
This is a Phase 1, randomized, open-label, 2-way crossover, pharmacokinetic study in adult patients with hematological malignancies eligible to receive either cyclophosphamide, doxorubicin, vincristine, and prednisone (CHOP) regimen or rituximab-CHOP (R-CHOP) regimen.

DETAILED DESCRIPTION:
Eligible patients will be randomized in a 1:1 ratio to one of 2 treatment cohorts (Cohorts A or B) in which the Marqibo formulation and the 1-vial VSLI-RTU formulation of vincristine are administered in a 2-way crossover design over 2 treatment cycles (21 days each):

* Cohort A: Marqibo formulation given at a dose of 2.25 mg/m2 with no dose cap during Cycle 1, and VSLI-RTU formulation given at 2.25 mg/m2 with no dose cap during Cycle 2.
* Cohort B: VSLI-RTU formulation given at a dose of 2.25 mg/m2 with no dose cap during Cycle 1 and Marqibo formulation given at 2.25 mg/m2 with no dose cap during Cycle 2.

Both formulations of vincristine sulfate LIPOSOME injection will be administered via a 60 (±10) minute IV infusion.

Blood samples for PK evaluation will be drawn at the following time points: immediately before infusion, 0.5 hour after the start of the infusion, 0.5 hour after the end of infusion (EOI), and 3, 8, 15, 24, 48, 72, and 96 hours post-EOI.

In addition to Marqibo or VSLI-RTU, all patients will receive standard doses (per institutional or regional guidelines) of cyclophosphamide, prednisone, and doxorubicin, (and rituximab if patient is on the R-CHOP regimen), on Day 1 and prednisone (or prednisolone if consistent with institutional or regional guidelines) on Days 2 to 5.

ELIGIBILITY:
Key Inclusion Criteria:

* Patient has a hematological malignancy and is eligible to receive CHOP or R-CHOP regimen.
* Patient must have adequate hematological, renal, and hepatic function as specified below within 30 days prior to the first dose of study treatment:
* Patient has a left ventricular ejection fraction ≥50% by multigated acquisition scan or echocardiogram within 30 days prior to the first dose of study treatment.

Key Exclusion Criteria:

* Patient has severe neurologic disorders (Grade 3 and above) including peripheral motor and sensory, central and autonomic neuropathy.
* Patient has a history of persistent active neurologic disorders including the demyelinating form of Charcot-Marie-Tooth syndrome, acquired demyelinating disorders, and other demyelinating conditions.
* Patient has used any investigational drugs, biologics, or devices within 30 days prior to study treatment or plans to use any of these during the course of the study.
* Patient has bowel obstruction, paralytic ileus, or uncontrolled chronic constipation.
* Patient has severe, active and uncontrolled hepatic disease or dysfunction.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2020-08-15 (Estimated); Primary Completion 2020-08-15 (Estimated); Study Completion 2020-10-15 (Estimated)

PRIMARY OUTCOMES:
PK analysis Area under the concentration time curve (AUC) | 6 weeks
  To evaluate the serum pharmacokinetics (PK) of the 1-vial VSLI-RTU formulation versus the current Marqibo 3-vial formulation for intravenous (IV) injection.

CONTACTS AND LOCATIONS:
Overall Officials: Wasim Khan, MD, Study Director — Acrotech Biopharma Inc.

IPD SHARING:
Plan to Share IPD: No